CLINICAL TRIAL: NCT00427791
Title: Phase II Randomized Study Evaluating the Addition of Rituximab to the Preparative Regimen of Etoposide and Total Body Irradiation in Acute Lymphoblastic Leukemia
Brief Title: Rituximab to the Preparative Regimen of Etoposide and Total Body Irradiation in Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0989
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Results first posted 2012-05-07 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2012-04

CONDITIONS: Leukemia
Keywords: Acute Lymphoblastic Leukemia; Leukemia; Total Body Irradiation; Etoposide; Rituximab; Rituxan; TBI; ALL
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Etoposide; Whole-Body Irradiation; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Etoposide + Total Body Irradiation + Rituximab (Experimental): Etoposide 60 mg/kg intravenous (IV) Daily Over 4 Hours for 1 Day + Total Body Irradiation (TBI) 3 Gy Daily for 4 Days + Rituximab 375 mg/m^2 IV Weekly Over 4-8 Hours for 4 Weeks
  Interventions: Drug: Etoposide; Radiation: Total Body Irradiation; Drug: Rituximab
- Etoposide + Total Body Irradiation (Experimental): Etoposide 60 mg/kg IV Daily Over 4 Hours for 1 Day + TBI 3 Gy Daily for 4 Days
  Interventions: Drug: Etoposide; Radiation: Total Body Irradiation

INTERVENTIONS:
Drug: Etoposide — 60 mg/kg IV Daily Over 4 Hours for 1 Day
Radiation: Total Body Irradiation — 3 Gy Daily for 4 Days
  Other Names: TBI
Drug: Rituximab — 375 mg/m^2 IV Weekly Over 4-8 Hours for 4 Weeks
  Other Names: Rituxan
  Arms: Etoposide + Total Body Irradiation + Rituximab

SUMMARY:
Primary Objective:

* To determine the progression free survival (PFS) of the preparative regimen rituximab, etoposide and total body irradiation (TBI), in patients with acute lymphoblastic leukemia (ALL) receiving allogeneic hematopoietic stem cell transplantation (SCT).

Secondary Objectives:

* To determine the effect of rituximab on the incidence of acute graft vs. host disease (GVHD).
* To determine the efficacy of adding imatinib mesylate post transplant in ALL patients with the t(9;22)(q34;q11) cytogenetic abnormality.
* To estimate the probability of molecular complete remission at one year for the described treatment approach as determined by serial minimal residual disease (MRD) monitoring.
* To determine the rate of GVHD, engraftment, toxicity, and overall survival (OS) for this treatment regimen.

DETAILED DESCRIPTION:
Disease relapse and GVHD are 2 factors that significantly impact survival in ALL patients who receive SCT. GVHD occurs when donor cells (graft) attack the stem cell recipient's (host's) cells. The term "acute" refers to the time it takes for the GVHD to appear after the transplant. This time frame is usually within the first 100 days after the transplant. GVHD occurs in up to 50% of patients who receive a transplant.

Etoposide is a traditional chemotherapy drug that is designed to interfere with the production of cancer cells at the DNA and RNA level. Total body irradiation (TBI) uses low level radiation to also interfere with the production of cancer cells at the DNA and RNA level. The combination of etoposide and TBI is a standard transplant conditioning therapy used for ALL patients. Rituximab is a monoclonal antibody that is designed to work against cells that express the antigen CD20. In addition, some studies suggest that it may decrease the risk of GVHD.

Before you can start treatment on this study, you will have what are called "screening tests". These tests will help the doctor decide if you are eligible to take part in the study. You will have a complete medical history and physical exam, including routine blood (2-3 teaspoons) and urine tests. You will have a chest x-ray, heart scan (echocardiogram or MUGA scan (Multi Gated Acquisition Scan)), lung function test, and a bone marrow biopsy with aspirate to evaluate the status of your disease before transplant. To collect a bone marrow biopsy and aspirate, an area of the hip or chest bone is numbed with anesthetic, and a small amount of bone marrow and bone is withdrawn through a large needle. A bone marrow core (a solid piece from the bone marrow) is also collected through a hollow needle inserted into the hip bone. Women who are able to have children must have a negative blood pregnancy test.

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the toss of a coin) to one of 2 treatment groups. Participants in one group will receive etoposide and TBI before their transplant. Participants in the other group will receive etoposide, TBI, and rituximab before their transplant. There is an equal chance of being assigned to either group. You will receive treatment on this study as an inpatient.

On the 1st day of hospitalization, you will receive fluids by vein through a central venous catheter (a plastic tube inserted into a large vein under your collar bone). You will receive TBI, once a day for the next 4 days. During TBI, you will lie flat on a table and receive radiation beams to all parts of the body, with shielding over certain parts of the body. On the following day, you will receive etoposide through the catheter over 4 hours. You will then have 2 days of rest, followed by your transplant of stem cells. The stem cells will be infused into your vein. The infusion can last from 30 minutes to several hours.

If you are assigned to the rituximab group, you will also receive rituximab once a week for 4 weeks by vein over 4-8 hours. The first dose will be given on the first day you receive etoposide. If you are receiving a mismatched-related allogeneic stem cell transplant or an unrelated allogeneic stem cell transplant, you will also receive Thymoglobulin by vein on the 3 days before the stem cell infusion. This is given to decrease the risk of GVHD and graft rejection in mismatched transplants.

In addition, you may receive a supportive care drug called palifermin (Kepivance®), which is a human keratinocyte growth factor (KGF) produced by recombinant DNA technology in E. coli. Its use has been shown to decrease mucositis resulting from high dose chemotherapy used in stem cell transplantation. You may receive palifermin for 3 days before starting radiation therapy, and for 2 days beginning on the day of your stem cell infusion. You may not receive palifermin but you will still receive transplant.

After you blood counts have normalized following your stem cell transplant, you will start taking imatinib mesylate by mouth only if your disease has the Philadelphia chromosome (Ph+ ALL). Approximately 25-30% of adults with ALL harbor the Philadelphia chromosome. You will take it once a day until 1 year after your transplant. Imatinib mesylate should be taken with a meal and a glass of water, preferably in the morning. The dose will be gradually increased as long as you don't experience severe side effects. If severe side effects occur, imatinib will be stopped, either temporarily or permanently.

You will receive several other medications to help the treatment work and to help decrease the risk of infections while your immune system is weak. Tacrolimus and methotrexate will be given to decrease the risk of GVHD. The tacrolimus will be started on the day before the transplant and will continue for up to 6 months. Tacrolimus is given by vein at first and then by mouth when you are able to eat. Methotrexate is given by vein on Days 1, 3, 6, and 11 after the transplant.

Sulfamethoxazole (Bactrim) or pentamidine will be given to fight bacteria. Bactrim is given by mouth when your blood counts are good. Pentamidine is given by vein when the counts are low. Acyclovir will be given at first by vein and then Valtrex (valacyclovir) will be given by mouth to decrease the risk of viral infections. Both of these will be given as per standard of care. Granulocyte colony-stimulating factor (G-CSF) will be given to help the new bone marrow grow. It is given as an injection under the skin after the transplant. It will continue until the white blood cells reach an acceptable level. These are all routine supportive medications used during bone marrow transplantation. Overall, some of these drugs will be given for as long as 6 months or possibly longer. Other medications may be necessary. If you are allergic to some of these drugs, changes will be made.

You will be in the hospital for about 3-4 weeks. You will have checkups every day until you are discharged from the hospital. You will then be seen in the outpatient clinic at least 3 times a week until your blood counts improve. You will be seen by your doctor at least every week until 100 days after the bone marrow transplant. You must stay in Houston during this time. After 100 days, you will be required to return to Houston every 3 months for tests and evaluation over the next 2 years. At these visits, you will have blood (about 2-3 teaspoons) collected for routine tests. You will also have a bone marrow biopsy.

Some participants may need to receive spinal taps with chemotherapy (methotrexate or cytarabine given through the spine) several times over the year after transplantation. This is only for patients with a previous clinical history of leukemic involvement of the brain or high risk of developing leukemia relapse in the brain. The spinal tap is performed in the clinic. If you are one of these participants, you will be given local anesthetic at the lower back site where a small needle will be inserted in the space between 2 spinal bones. A small amount of fluid that bathes the brain (cerebrospinal fluid) will be removed for testing, and a small amount of chemotherapy will be given.

This is an investigational study. The FDA has approved all of the drugs used in this study for use in stem cell transplantation. However, their use together in this study is experimental. Up to 80 patients will take part in this study. All will be enrolled at UT MD Anderson Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy-proven ALL in remission or relapse.
* Adequate renal function, as defined by estimated serum creatinine clearance >50 ml/min and/or serum creatinine <1.8 mg/dL.
* Adequate hepatic function, as defined by aspartate aminotransferase (AST) or serum glutamic oxaloacetic transaminase (SGOT) <3 * upper limit of normal; serum bilirubin and alkaline phosphatase <2 * upper limit of normal, or considered not clinically significant.
* Adequate pulmonary function with Forced Expiratory Volume in One Second (FEV1), forced vital capacity (FVC) and Carbon Monoxide Diffusing Capacity (DLCO) at least 45% of expected corrected for hemoglobin.
* Adequate cardiac function with left ventricular ejection fraction at least 45%. No uncontrolled arrhythmias or symptomatic cardiac disease.
* Zubrod performance status <2.
* Patients must have a related, genotypically human leukocyte antigens (HLA) identical donor, or they must have a related or unrelated donor who is at least a 9/10 HLA match by high resolution typing.
* Female patient must not be pregnant and have negative pregnancy test.
* Patient and donor should be willing to participate in the study by providing written consent.

Exclusion Criteria:

* Patients with unresolved grade 3 or greater non-hematologic toxicity from previous therapy. Patients with grade 2 toxicity will be eligible at the discretion of the principal investigator (PI).
* Patients with active central nervous system (CNS) disease.
* Evidence of acute or chronic active hepatitis or cirrhosis.
* Uncontrolled infection, including Human immunodeficiency virus (HIV) or Human T-lymphotropic virus Type I (HTLV-1) infection.
* Patients greater than 60 years-old.
* Prior autologous or allogeneic hematopoietic stem cell transplant.

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2005-07; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Partow Kebriaei, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: July 05, 2005 to August 08, 2008. All participants were enrolled at UT MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | Etoposide + Total Body Irradiation + Rituximab | Etoposide + Total Body Irradiation
Started | 10 | 13
Completed | 10 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Etoposide + Total Body Irradiation + Rituximab | Etoposide + Total Body Irradiation | Total
Number analyzed (Participants) | 10 | 13 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 10 | 12 | 22
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 7 | 9 | 16
Region of Enrollment [Number; unit: participants]
  United States | 10 | 13 | 23

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Time from randomization to first progression or death, whichever comes first, measured in months.
Time Frame: 2 Years post transplant or until disease progression or death
Population: Analysis was by protocol. Participants were randomized between Etoposide + Total body irradiation and Etoposide + Total body irradiation + Rituximab using a Bayesian adaptive algorithm.
Measure: Median (Standard Deviation); unit: Months
Arm/Group | Etoposide + Total Body Irradiation + Rituximab | Etoposide + Total Body Irradiation
Number analyzed (Participants) | 10 | 13
Months | 4.3 (0.95) [1 to 10] | 14.5 (0.95)

2. Secondary Outcome: Number of Participants With Incidence of Acute Graft Versus Host Disease During First 100 Days
Description: Number of participants with incidence of acute graft versus host disease (aGVHD) during first 100 days following transplant.
Time Frame: During the first 100 days following transplant
Population: Analysis was by protocol.
Measure: Number; unit: participants
Arm/Group | Etoposide + Total Body Irradiation + Rituximab | Etoposide + Total Body Irradiation
Number analyzed (Participants) | 10 | 13
participants | 5 | 9

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Etoposide + Total Body Irradiation + Rituximab | Etoposide + Total Body Irradiation
Serious Adverse Events (participants affected / at risk) | 10/10 | 2/13
Other Adverse Events (participants affected / at risk) | 10/10 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etoposide + Total Body Irradiation + Rituximab (N=10) | Etoposide + Total Body Irradiation (N=13)
Hypertension (Cardiac disorders) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis (Gastrointestinal disorders) | 5 (5) | 1 (1)
GI Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Transiminitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Venous occlusive disease (Hepatobiliary disorders) | 1 (1) | 0 (0)
Other (Pain) (Nervous system disorders) | 2 (2) | 0 (0)
Pneumonitis (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etoposide + Total Body Irradiation + Rituximab (N=10) | Etoposide + Total Body Irradiation (N=13)
Edema (Cardiac disorders) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 2 (2) | 3 (3)
Lethargy (General disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 9 (9) | 9 (9)
Mucositis (Gastrointestinal disorders) | 3 (3) | 9 (9)
Nausea (Gastrointestinal disorders) | 6 (6) | 7 (7)
GvHD (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 5 (5) | 9 (9)
Hemorrhagic cystitis (Renal and urinary disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 6 (6) | 5 (5)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Bone pain (General disorders) | 0 (0) | 2 (2)
Neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Neurologic (General disorders) | 2 (2) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes